CLINICAL TRIAL: NCT06297122
Title: Severe Group A Streptococcus Infections in Children During the COVID-19 Pandemic: an Interrupted Time-series Analysis in Paris, France, 2018-2023
Brief Title: Severe Group A Streptococcus Infections in Paris, France, 2018-2023
Acronym: IGASI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240002
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Invasive Group A Beta-Haemolytic Streptococcal Disease
Keywords: Group A Streptococcus (GAS) infection; Pediatric severe GAS infections; GAS infection incidence; COVID-19 pandemic; Time-series analysis
MeSH Terms: conditions — Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: All consecutive children under the age of 18 years with community-acquired or healthcare-associated severe Group A Streptococcus (GAS) infections admitted to Necker hospital between January 1, 2018, and December 31, 2023. Among GAS infections, invasive and probable invasive GAS illnesses will be distinguish.
  "Invasive GAS" infection will be defined as: isolation by culture or polymerase chain reaction of GAS from a normally sterile site; or isolation of GAS from a sterile or non-sterile site accompanied by necrotizing fasciitis or streptococcal toxic shock syndrome.
  "Probable invasive" GAS will be defined as acute infections with GAS isolated from a non-sterile site, which includes sputum, otorhinolaryngology surgical specimens (mastoiditis, ethmoiditis, pharyngeal abscess) accompanied with one or more of the following severity criteria:intravenous antibiotics;surgery; and/or admission to the pediatric intensive care unit.
  Interventions: Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file (electronic health record). The identification of eligible cases will be conducted through an examination of the hospital's electronic microbiology database. Subsequently, the complete hospital record(s) of each patient will be used to extract a pre-defined set of variables required for data analysis.

SUMMARY:
Streptococcus pyogenes, commonly referred to as Group A Streptococcus (GAS), has the ability to induce a diverse range of illnesses.

In several European countries and the United States, a notable surge in invasive GAS (iGAS) infections has been documented since mid-2022. This sharp increase contrasts with the gradual rise in iGAS incidence observed among children over the past three decades. As demonstrated for several viral infections, the recent upturn in iGAS infections is potentially linked to the relaxation of mitigation measures implemented during the COVID-19 pandemic, such as face mask usage and school closures.

Since November 2022, concerns have been raised by French public health authorities regarding the rise in levels of iGAS infections, and an unexpected increase in pediatric severe GAS infections was reported in a French single-center study. However, this study ended in December 2022 and could only explore short-term trends. The Necker - Enfants malades Hospital in Paris, France, represents an excellent opportunity to examine the impact of the COVID-19 pandemic and the associated non-pharmaceutical interventions on the incidence of severe GAS infections, during, and after the pandemic.

This study aims to investigate trends of severe GAS infection incidence in children in the Paris area over the course of the COVID-19 pandemic.

DETAILED DESCRIPTION:
Streptococcus pyogenes, commonly referred to as Group A Streptococcus (GAS), has the ability to induce a diverse range of illnesses. In primary care, acute pharyngitis, commonly known as 'strep throat', is the predominant form of GAS infection. Other commonly encountered non-invasive GAS infections encompass impetigo, scarlet fever, perianal infections, and paronychia. GAS may also cause rarer yet severe conditions such as streptococcal toxic shock syndrome, pneumonia with pleural empyema, and septic shock; most severe GAS infections can even be life-threatening.

In several European countries and the United States, a notable surge in invasive GAS (iGAS) infections has been documented since mid-2022. This sharp increase contrasts with the gradual rise in iGAS incidence observed among children over the past three decades. As demonstrated for several viral infections, the recent upturn in iGAS infections is potentially linked to the relaxation of mitigation measures implemented during the COVID-19 pandemic, such as face mask usage and school closures. Non-pharmaceutical interventions and behavioral changes during the COVID-19 pandemic modified the spread of SARS-CoV-2 and several respiratory pathogens, including GAS. Reduced exposure to endemic infectious agents may have created an immunity gap, leading to unexpected epidemics of viral and bacterial infections after non-pharmaceutical interventions were relaxed.

Since November 2022, concerns have been raised by French public health authorities regarding the rise in levels of iGAS infections, and an unexpected increase in pediatric severe GAS infections was reported in a French single-center study. However, this study ended in December 2022 and could only explore short-term trends. The Necker - Enfants malades Hospital in Paris, France, represents an excellent opportunity to examine the impact of the COVID-19 pandemic and the associated non-pharmaceutical interventions on the incidence of severe GAS infections, during, and after the pandemic. This tertiary care university hospital is located in a densely populated region and has various specialized departments involved in the management of severe infections, including pediatric intensive care units (PICU), orthopedics, pulmonology, otolaryngology, dermatology, infectious diseases, and microbiology.

This study aims to investigate trends of severe GAS infection incidence in children in the Paris area over the course of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 18 years.
* Admitted to Necker-Enfants Malades hospital for community-acquired or healthcare-associated severe Group A Streptococcus (GAS) infections between January 1, 2018, and December 31, 2023.
* Severe GAS infections comprises "invasive" and "probable invasive" GAS illnesses.

"Invasive" GAS infection will be defined as:

* isolation by culture or polymerase chain reaction (PCR) of GAS from a normally sterile site (e.g., blood, pleural fluid, cerebrospinal fluid, joint fluid, bone, bronchoalveolar lavage fluid); or
* isolation of GAS from a sterile or non-sterile site accompanied by necrotizing fasciitis or streptococcal toxic shock syndrome.

"Probable invasive" GAS will be defined as acute infections with GAS isolated from a non-sterile site, which includes sputum, otorhinolaryngology surgical specimens (mastoiditis, ethmoiditis, pharyngeal abscess) accompanied with one or more of the following severity criteria:

* intravenous (IV) antibiotics;
* surgery; and/or
* admission to the PICU.

Exclusion Criteria:

* Non-severe GAS infection, such as acute otitis media with otorrhea, pharyngitis, scarlet fever, GAS skin carriage.
* GAS identified on minor/superficial skin lesions.
* Otolaryngology infections (e.g., parapharyngeal abscess) that do not require IV antibiotics, surgery, or PICU admission.
* Opposition to the use of routine data.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutive children under the age of 18 years with community-acquired or healthcare-associated severe Group A Streptococcus (GAS) infections admitted to Necker-Enfants Malades hospital between January 1, 2018, and December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Monthly incidence of severe Group A Streptococcus (GAS) infections per 1000 pediatric hospital admissions | 6 years
  The monthly incidence of severe group A streptococcal infections per 1000 pediatric hospital admissions.
  Two specific breakpoints in the data will be used: March 2020, marking the first lockdown, and March 2022, marking the point when mask-wearing in schools was no longer mandatory. This will allow to define four distinct periods for analysis:
  * January 2018 to March 2020 (pre-pandemic period),
  * April 2020 to March 2022 (early pandemic period),
  * April 2022 to September 2023 (late pandemic period), and
  * May 2023 to December 2023 (post pandemic period).

SECONDARY OUTCOMES:
Age of children age with group A Streptococcus (GAS) infections | 6 years
  Description of possible changes in characteristics of severe Group A Streptococcus (GAS) infections between the defined periods, in terms of children age (in years).
Proportion of children needing surgical intervention for the management of GAS infection | 6 years
  Description of possible changes in characteristics of severe Group A Streptococcus (GAS) infections between the defined periods, in terms of proportion of children needing surgical intervention for the management of GAS infection (in %).
Proportion of cases admitted in the PICU for GAS infection | 6 years
  Description of possible changes in characteristics of severe Group A Streptococcus (GAS) infections between the defined periods, in terms of proportion of cases admitted in the PICU (in %).
Proportion of deaths from GAS infection | 6 years
  Description of possible changes in characteristics of severe Group A Streptococcus (GAS) infections between the defined periods, in terms of proportion of deaths (in %).
Hospital length of stay for the management of GAS infection | 6 years
  Description of possible changes in characteristics of severe Group A Streptococcus (GAS) infections between the defined periods, in terms o fhospital length of stay (in days).
Distribution of infection type of GAS infection | 6 years
  Description of possible changes in characteristics of severe Group A Streptococcus (GAS) infections between the defined periods, in terms of distribution of infection type (in %). For example arthritis, empyema, pharyngeal abscess, isolated bacteremia. In the event of multiple diagnoses, the most serious will be kept.
Proportion of healthcare-associated infections during the management of GAS infection | 6 years
  Description of possible changes in characteristics of severe Group A Streptococcus (GAS) infections between the defined periods, in terms of proportion of healthcare-associated infections (in %).

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Cohen, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Alix Flamant, M.D., Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flamant A, Faury H, Luscan R, Couloigner V, Pouletty M, Bustarret O, Chappuy H, Gaume M, Drummond D, Pinhas Y, Toubiana J, Ferroni A, Cohen JF. Severe Group A Streptococcus Infections in Children During and After the COVID-19 Pandemic: An Interrupted Time-series Analysis in Paris, France, 2018-2023. Pediatr Infect Dis J. 2025 Oct 1;44(10):973-978. doi: 10.1097/INF.0000000000004872. Epub 2025 May 28. PMID 40440703